CLINICAL TRIAL: NCT00848185
Title: Differential Regulation of VEGF, Cadherin and Angiopietin 2 by Trigger Oocyte Maturation With GnRHa vs hCG in Donors: Try to Explain the Lower OHSS Incidence
Brief Title: Differential Regulation of VEGF, Cadherin, Angiopietin 2 by Trigger Oocyte Maturation With GnRHa vs hCG in Donors
Status: Completed | Type: Observational
Sponsor: IVI Madrid (Other)
Responsible Party: Principal Investigator, Juan A Garcia-Velasco, MD PhD, IVI Madrid
Other Study IDs: IVIMAD-MC-10-2008-01
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2017-04-17 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-04

CONDITIONS: Vascular Endothelial Growth Factor Overexpression
Keywords: VEGF; Trigger; OHSS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — follicular fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Antagonist-hCG for triggering: Protocol with antagonist and hCG to trigger oocyte maturation
- Antagonist-aGnRH for triggering: Protocol with antagonist and 0,2 mg triptorelin to trigger oocyte maturation
- Long protocol-hCG for triggering: Long Protocol and hCG to trigger oocyte maturation

SUMMARY:
Introduction OHSS still remains a complication of assisted reproduction treatments. hCG administration to trigger final oocyte maturation will release vascular mediators, being VEGF and other proteins such as VE-Cadherin or Angiopoietin- 2. It has been shown that replacing hCG by GnRH agonists will induce a very short endogenous LH peak, potent enough to induce final oocyte maturation but no OHSS will develop. The investigators examined VEGF, VE-Cadherin and Angiopoietin-2 modulation by hCG as well as GnRH agonists in oocyte donors undergoing controlled ovarian stimulation.

DETAILED DESCRIPTION:
Material and Methods Between June and December of 2008 we evaluated 90 egg donors. They underwent COH with 150 IU rFSH as starting dose, we separated them in 3 groups (n:30 each): Groups 1 and 2 received a 0.25mg daily dose of GnRH antagonist when a follicle 14mm in diameter was observed. hCG 250g was given to group 1 while group 2 received triptorelin 0.2mg when leading two follicles were 17mm. Group 3 was stimulated with standard long protocol, hCG was given following similar criteria.

Blood was collected the day of hCG/aGnRH administration as well as the day of egg retrieval, and follicular fluid from the first two mature follicles was also frozen. We collected granulosa cells (GC) of 10 patients of each group as well Levels of VEGF, sVE-Cadherin an Angiopietin 2 were determined by ELISA in serum and in follicular fluid.

Results were analyzed via ANOVA.Data are expressed as mean± SEM. A significant difference was defined as p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Donors

Exclusion Criteria:

* Important diseases

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: oocyte Donors
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Antagonist Trigger With aGnRH: Protocol with antagonist and 0,2 mg triptorelin to trigger oocyte maturation
- Antagonist Trigger With hCG: Protocol with antagonist and hCG to trigger oocyte maturation
- Long Protocol hCG: Long Protocol with hCG to trigger oocyte maturation
Period: Overall Study
Arm/Group | Antagonist Trigger With aGnRH | Antagonist Trigger With hCG | Long Protocol hCG
Started | 32 | 32 | 32
Completed | 32 | 32 | 32
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: * Age between 18 and 35 years and previous pregnancy
  * Regular menstrual cycles (between 25 and 35 days)
  * Normal karyotype
  * Body massindex between 18 and 25 kg/m2
  * Negative serology for VHB, VHC and HIV
  * Normal cervical cytology in the past year, and a vaginal ultrasound without evidence of any pathologic conditions
Groups:
- Antagonist-hCG to Trigger: Protocol with antagonist and hCG to trigger oocyte maturation
- Antagonist-aGnRH to Trigger: Protocol with antagonist and 0.2 mg triptorelin to trigger oocyte maturation
- Long Protocol-hCG: Long Protocol and hCG to trigger oocyte maturation
- Total: Total of all reporting groups
Arm/Group | Antagonist-hCG to Trigger | Antagonist-aGnRH to Trigger | Long Protocol-hCG | Total
Number analyzed (Participants) | 32 | 32 | 32 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 32 | 32 | 32 | 96
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.2 (3.5) | 23.7 (3.9) | 24.5 (3.7) | 25.1 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 32 | 32 | 96
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — The donors were recruit for the clinic
  participants
    Spain | 32 | 32 | 32 | 96

OUTCOME MEASURES:

1. Primary Outcome: VEGF Protein and mRNA Levels
Description: VEGF concentration in follicular fluid and VEGF mRNA expression in granulosa cells from patients who received either GnRH agonist instead of hCG
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: pg/ml
Groups:
- Antagonist-hCG Levels of VEGF: Levels of VEGF in folicular fluid of patients with antagonist protocol anf hCG for triggering
- Antagonist-aGnRH Levels of VEGF: Levels of VEGF in folicular fluid of patients with antagonist protocol and aGnRH for triggering
- Long Protocol- hCG: Levels of VEGF in folicular fluid of patients with long protocol anf hCG for triggering
Arm/Group | Antagonist-hCG Levels of VEGF | Antagonist-aGnRH Levels of VEGF | Long Protocol- hCG
Number analyzed (Participants) | 32 | 32 | 32
pg/ml | 1395 (284) | 1069 (354) | 1666 (55)
Statistical Analysis 1: Comparison: Antagonist-hCG Levels of VEGF vs Antagonist-aGnRH Levels of VEGF vs Long Protocol- hCG; ANOVA for three groups; Test type: Superiority or Other; p < 0.001, ANOVA

ADVERSE EVENTS:
Groups:
- GnRH Antagonist - hCG Trigger: GnRH antagonist protocol and hCG trigger
- GnRH Antagonist Triptorelin Trigger: GnRH antagonist protocol and triptorelin trigger
- Long Protocol - hCG Trigger: Long protocol and hCG trigger as control
Arm/Group | GnRH Antagonist - hCG Trigger | GnRH Antagonist Triptorelin Trigger | Long Protocol - hCG Trigger
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No